CLINICAL TRIAL: NCT07151586
Title: A Phase 2, Multicenter, Randomized, Open-label Trial Assessing Sacituzumab-govitecan and Trastuzumab-deruxtecan Combinations in an Alternating Regimen for Patients With Metastatic or Locally Advanced HER2-low Triple-negative Breast Cancer
Brief Title: Testing Two Different Drugs (Sacituzumab-govitecan and Trastuzumab-deruxtecan) Combinations Prescribed in an Alterning Pattern to Patients With Metastatic or Locally Advanced Triple-negative Breast Cancer
Acronym: ALTER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-BCG-2503; 2025-521909-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Triple Negative Breast Neoplasms; Neoplasm Metastasis; HER 2 Low-expressing Breast Cancer
Keywords: Antibody-drug conjugates; HER2-low; Triple Negative Breast Cancer; Locally Advanced Breast Cancer; HER2-negative; Metastatic Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm Metastasis; Breast Neoplasms | interventions — sacituzumab govitecan; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacituzumab-Govitecan and Trastuzumab-deruxtecan in alternating shema (Experimental): Patients will receive either SG and T-DXd in an upfront alternating schema: two cycles of SG, followed by two cycles of T-DXd, then two cycles of SG, and so on, until RECIST 1.1-defined disease progression, unless there is unacceptable toxicity, withdrawal of consent or end of study.
  Interventions: Drug: Sacituzumab Govitecan / Trastuzumab Deruxtecan
- Sacituzumab-Govitecan alone (Active Comparator): Patient will receive Sacituzumab-Govitecan 1(monotherapy) until RECIST 1.1-defined disease progression, unless there is unacceptable toxicity, withdrawal of consent or end of study
  Interventions: Drug: Sacituzumab Govitecan / Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Sacituzumab Govitecan / Trastuzumab Deruxtecan — Sacituzumab govitecan is administered intravenously at a dose of 10 mg/kg on Day 1 and Day 8 of each 3-week cycle. In this study, patients receive two cycles of sacituzumab govitecan followed by two cycles of trastuzumab deruxtecan, alternating throughout the study.
  Trastuzumab deruxtecan is administered intravenously at a dose of 5.4 mg/kg on Day 1 of each 3-week cycle. In this study, patients receive two cycles of trastuzumab deruxtecan followed by two cycles of sacituzumab govitecan, alternating throughout the study.
  Both Treatment are continued until disease progression as defined by RECIST 1.1, unacceptable toxicity, withdrawal of consent, or the end of the study.
  Other Names: Trodelvy; Enhertu

SUMMARY:
This is a phase II, multicentre, open-label, randomised controlled trial (patients are randomly assigned to one treatment arm or the other) evaluating two treatment strategies (sacituzumab govitecan and trastuzumab deruxtecan in an alternative schema or sacituzumab govitecan alone) in patients with locally advanced or metastatic triple-negative breast cancer.

The goal is to answer the question: Does alternating sacituzumab goveitecan (SG) and trastuzumab deruxtecan (T-DXd) improve survival in patients with HER2-low metastatic triple-negative breast cancer compared to continuing treatment with SG alone?

DETAILED DESCRIPTION:
Patients with locally advanced or metastatic triple-negative breast cancer (mTNBC) have poor survival outcomes

Among mTNBC, about 40% of tumors have a low expression of HER2 (HER2-low; defined as IHC 2+/ISH or IHC 1+). Two antibody-drug conjugates (ADCs) have been approved for HER2-low mTNBC: sacituzumab govitecan (SG) and trastuzumab deruxtecan (T-DXd) that target TROP2 and HER2 at the tumor cell surface, respectively. Each of these ADCs, used as monotherapy, outperformed conventional chemotherapy according to the ASCENT and DESTINY-Breast 04 trials and thereby have become the new second or third line standard of care for HER2-low mTNBC. However, as with other types of treatments, resistance is inescapable mostly due to intra-tumor heterogeneity. In the case of ADCs, resistance mechanisms involve changes in tumor antigen expression, ADC intracellular uptake and processing, and efflux of the ADC cytotoxic payload. Consequently, SG and T-DXd are used sequentially after progression even though the most effective sequence has so far been scarcely investigated and remains to be established

The ASCENT trial was designed to compare the efficacy of SG with chemotherapy in patients with mTNBC and reported significantly greater progression-free and overall survival compared with the physician's choice of chemotherapy. On the other hand, the DESTINY-Breast-04 compared the efficacy of T-DXd with chemotherapy but included just 63 patients with HER2-low mTNBC. Despite a significantly longer progression-free and overall survival were observed compared with the physician's choice of chemotherapy the efficacy analysis of T-DXd in this subpopulation was not a prespecified endpoint of the trial. Even though, collectively these results have contributed to a treatment paradigm shift for mTNBC, the superiority to chemotherapy can only be formally claimed for SG in mTNBC patients and for T-DXd in HER2-low metastatic breast cancer patients

We hypothesize that an upfront alternating SG and T-DXd regimen would have a greater antitumor effect compared with their prescription at progression while limiting the emergence of drug resistance. Hence, the ALTER trial aims to compare the efficacy and safety of an upfront alternating SG and T-DXd regimen with SG alone in HER2-low mTNBC patients

ELIGIBILITY:
Inclusion Criteria:

* Patient must have signed a written informed consent prior to any trial specific procedures. (Note : When the patient is physically unable to give his/her written consent, a impartial witness of their choice, independent from the investigator or the sponsor, can confirm in signing the patient's consent)
* Men or women ≥ 18 years of age
* Histologically confirmed metastatic or locally advanced and unresectable triple-negative breast cancer, meeting both of the following criteria by local testing:

HER2-low breast cancer, defined as either immunohistochemistry (IHC) 2+ / in situ hybridization (ISH)-negative or IHC 1+ (ISH-negative or untested), on either the primary or any metastatic site

Estrogen receptor (ER) expression <10% and progesterone receptor (PR) expression <10% (Note: In case of bilateral breast cancer, participation in the study is permitted as long as both tumours correspond to a triple-negative breast cancer meeting the above criteria)

* Patient eligible to receive sacituzumab-govitecan and T-Dxd according to their indication
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Women of childbearing potential and male patients must agree to use adequate contraception for the duration of trial participation and up to 7 months after completing treatment for women and up to 4 months for men.

A woman is considered to be of childbearing potential if she is not postmenopausal or has not undergone hysterectomy. Postmenopausal is defined as any of the following:

Age ≥ 60 years Age < 60 years and ≥ 12 continuous months of amenorrhea with no identified cause other than menopause Surgical sterilization (bilateral oophorectomy)

- Adequate organ and bone marrow function within 28 days before enrollment. The most recent results available must be used for all parameters below:

Hemoglobin ≥ 9 g/dL. Red blood cell transfusion is not allowed within 1 week prior to screening assessment

Absolute neutrophil count (ANC) ≥ 1,500/mm³. Granulocyte-colony stimulating factor (G-CSF) administration is not allowed within 1 week prior to screening assessment

Platelet count ≥ 100,000/mm³. Platelet transfusion is not allowed within 1 week prior to registration

Total bilirubin ≤ 1.5 × upper limit of normal (ULN) if no liver metastases, or < 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastasis at baseline

Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN, or < 5 × ULN in patients with liver metastasis

Serum albumin ≥ 2.5 g/dL

Creatinine clearance (CrCl) ≥ 30 mL/min, calculated using the Cockcroft-Gault equation: CrCl (mL/min) = [(140 - age in years) × weight in kg] / [72 × serum creatinine in mg/dL] (× 0.85 for females)

* Adequate cardiac function, defined as a left ventricular ejection fraction ≥ 55% estimated by echocardiogram or multigated acquisition scintigraphy
* Women of childbearing potential must have a negative serum or urine pregnancy test done within 7 days before randomization
* Affiliated to the French Social Security System (or equivalent)
* Patient willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.

Exclusion Criteria:

* Patient previously treated with any ADC targeting HER2 or TROP2
* Patient with uncontrolled or significant cardiovascular disease
* Patients with brain metastases (BM) except for asymptomatic treated BM not requiring ongoing corticosteroid treatment with stable lesions on baseline/screening brain MRI. Patients who require treatment of brain metastases are eligible after 14 days post surgery or radiation, if felt to be clinically stable and not requiring ongoing corticosteroid treatment
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, or current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening
* Any medical history or condition that per protocol or in the opinion of the investigator is incompatible with the study
* Patients with known allergy or severe hypersensitivity to any of the trial drugs or their excipients
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may cause misleading study interpretation or prevent completion of study procedures and followup examinations
* Patients with any other disease or illness that requires hospitalisation or is incompatible with the trial treatment are not eligible
* Patients enrolled in another therapeutic trial within 30 days of inclusion
* Pregnant or breast-feeding women at the time of randomization or intention to become pregnant during the study and up to 7 months after treatment
* Person deprived of their liberty or under protective custody or guardianship
* Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, up to 4 years.
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | Time from randomization to disease progression, up to 4 years.
  Clinical Benefit Rate is defined as the percentage of patients with complete response (CR), partial response (PR), or stable disease (SD)for at least 24 weeks, as assessed by RECIST 1.1
Objective response rate (ORR) | Time from randomization to disease progression, up to 4 years.
  The objective response rate is defined as the percentage of patients with a complete response (CR) or a partial response (PR) as assessed by RECIST 1.1
Progression-free survival (PFS), | From randomization to disease progression or death, up to 4 years.
  The progression-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.
Quality-Adjusted progression free survival (QA-PFS) | From randomization to disease progression or death, up to 4 years.
  Quality-Adjusted progression free survival is calculated as the product of the progression free survival function and the overall health utility index EQ-5D-5L.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From first dose through 30 days after the last dose of study treatment
  Frequency and severity of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs), graded per NCI-CTCAE v5.0. The proportion of patients with treatment discontinuations, interruptions, or dose reductions due to adverse events will also be reported
Quality of Life questionnaire - EORTC QLQ-C30 | Baseline to Week 24
  Mean change from baseline in the EORTC QLQ-C30 Global Health Status/Quality of Life (GHS/QoL) score at Week 24. The QLQ-C30 is a 30-item questionnaire scored according to the EORTC scoring manual on 0-100 scales; higher GHS/QoL scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre TASSIN DE NONNEVILLE, Study Chair — Institut Paoli-Calmettes; François BERTUCCI, Study Chair — Institut Paoli-Calmettes
Locations (2):
- France (2):
  - institut Paoli calmette, Marseille
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.